CLINICAL TRIAL: NCT05155956
Title: Cerebral Hemodynamics and Microemboli During Placement of Relay®Branch Thoracic Stent-Graft System
Acronym: CHaMP
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: Bolton Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 850188
Record Dates: First submitted 2021-11-30; First posted 2021-12-14 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Thoracic Aortic Aneurysm; Thoracic Aortic Dissection; Microemboli
MeSH Terms: conditions — Aortic Aneurysm, Thoracic; Dissection, Thoracic Aorta | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: transcranial Doppler ultrasonography (TCD) — Transcranial Doppler (TCD) is a non-invasive ultrasound-based technique that facilitates insonation of the cerebral arteries. TCD probe design enables continuous monitoring of cerebral blood flow velocity (CBFv). TCD has a variety of clinical applications, including intraoperative monitoring for detection of microemboli. The TCD probe can be comfortably secured to the patient's head by a headframe in order to maintain continuous vessel insonation. Microembolic signals (MES) can be reliably detected based on standard criteria:
  1. Brief in duration (<300msec)
  2. High intensity (amplitude >3 dB above background)
  3. Unidirectional
  4. Audible chirp or snap
  Further, CBFv monitoring during may inform flow perturbations that occur during cardiac or vascular manipulations.

SUMMARY:
This is an observational cohort study addressing the incidence of cerebral microemboli and alterations of cerebral hemodynamic physiology of the Relay®Branch thoracic stent-graft system.

DETAILED DESCRIPTION:
This study is a prospective multi-center observational study. Eligible patients will be enrolled in RelayBranch (NCT03214601). Participating centers must have capabilities of performing intra-operative TCD monitoring and post-operative TCD monitoring. If sites have performed TCD microembolic monitoring during previous RelayBranch procedures, we will also incorporate these data in our analysis. The primary objective is to assess the number and timing of cerebral microemboli during Relay®Branch thoracic stent-graft deployment, to identify the highest risk portions of the procedure. Secondary objectives include: correlate procedural microembolic burden with neuroimaging and clinical outcome; quantify post-operative microemboli, correlating with neuroimaging and clinical outcome; and quantify the changes in cerebral blood flow and cerebral autoregulation that happens during critical procedural epochs, correlating with neuroimaging and clinical outcome.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in NCT03214601 based on presence of a thoracic aortic aneurysm, penetrating atherosclerotic ulcer, or chronic type B dissection that would require coverage of the brachiocephalic trunk and/or left carotid if a non-branching endograft were implanted Advanced heart failure with plan to treat with LVAD
* At least 18 years of age
* Patients enrolled prospectively must sign the informed consent form
* If patients underwent TCD monitoring during a previous RelayBranch procedure as part of routine clinical care, we will also incorporate their data in our analysis

Exclusion Criteria:

* Skull defect or skull surgery that will preclude monitoring
* Known lack of TCD temporal acoustic window (if had TCD in past)
* Expected surgical position will preclude access to the patient's head for monitoring

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 20 subjects will be enrolled at multiple participating centers. All eligible subjects will be identified based on enrollment in RelayBranch (NCT03214601) or in their hum. We anticipate enrollment will be complete within 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2021-12-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
number of intra-operative cerebral microemboli | during RelayBranch procedure
  TCD

SECONDARY OUTCOMES:
Post-operative microemboli (seen on post-op day 1 study) | post-op day 1
  TCD
Change in CBFv | intra-op and post-op day 1
  TCD
Change in cerebral autoregulation | intra-op and post-op day 1
  TCD

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Messe, MD, Principal Investigator — University of Pennsylvania
Locations (2):
- United States (2):
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Penn Presbyterian Medical Center, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Undecided